CLINICAL TRIAL: NCT06518681
Title: Prospective Clinical Trial Evaluating the Safety and Efficacy of Prosthetic Polymer Heart Valves for the Treatment of Aortic Valve Disease
Brief Title: Evaluating the Safety and Efficacy of Prosthetic Polymer Heart Valves for the Treatment of Aortic Valve Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Hearthill Medical Technology Co.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PoliaValve-SA-01
Record Dates: First submitted 2024-06-04; First posted 2024-07-24 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Regurgitation
Keywords: Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases; Ventricular Outflow Obstruction; Aortic Valve Stenosis; Aortic Valve Disease; Aortic Valve Regurgitation
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases; Ventricular Outflow Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PoliaValve (Aortic) (Experimental): Patients receiving the PoliaValve (Aortic) from HearrHill Medical
  Interventions: Device: PoliaValve (Aortic)

INTERVENTIONS:
Device: PoliaValve (Aortic) — Aortic Valve Replacement

SUMMARY:
The purpose of this study is to conduct the initial clinical investigation of the HeartHill Medical's polymer aortic valve, namely PoliaVavle，to collect evidence on the device's safety and performance.

DETAILED DESCRIPTION:
The polymer aortic valve, PoliaValve, from HeartHIll Medical, is indicated as a replacement for patients with severe aortic valve disease, including severe aortic stenosis, severe aortic regurgitation, or both. These patients will be included in the study after systematic assessment that the subjects meet the criteria for inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following conditions:

1. Subjects are ≥60 years old;
2. The subjects understand the nature and purpose of the research, voluntarily participate and sign the informed consent form, comply with the trial requirements, are willing to cooperate with surgical treatment and follow-up, and agree to relevant follow-up interviews and examinations;
3. The subject is diagnosed with severe aortic stenosis and/or regurgitation (or insufficiency) through echocardiography;
4. According to the 2020 ACC/AHA management guidelines for patients with valvular heart disease, the subject meets the indications for aortic valve replacement surgery and the preoperative assessment recommends surgical aortic valve replacement.

Exclusion Criteria:

Subjects must not meet any of the following conditions:

1. Other valve diseases with indications for surgery, such as severe mitral regurgitation, severe tricuspid regurgitation, moderate or above mitral stenosis, etc. require combined valve replacement, or had aortic valve surgery in the past;
2. Other serious cardiovascular diseases with indications for surgery, such as Stanford type A aortic dissection, aortic sinus aneurysm (sinus diameter >5.0cm), hypertrophic obstructive cardiomyopathy, diffuse three-vessel coronary artery disease , end-stage heart failure while simultaneously placing a left ventricular assist device, etc.;
3. End-stage heart failure that is expected to be irreversible by aortic valve surgery, such as severe left ventricular dysfunction with LVEF <25%, or severe heart failure that cannot be corrected, or severe pulmonary hypertension assessed by right heart catheterization, predict postoperative plans Perform Impella, IABP or left ventricular assist within the hospital;
4. Decompensated heart failure, cardiogenic shock, malignant arrhythmia, etc. that require mechanical circulatory assistance, mechanical ventilation or emergency surgery before surgery;
5. Active endocarditis or vegetations on the heart within 3 months;
6. History of severe acute myocardial infarction or cerebrovascular accident within 3 months (excluding lacunar infarction);
7. Those with severe renal insufficiency (GFR <30mL/min) or end-stage renal disease requiring long-term dialysis;
8. Liver dysfunction or gastrointestinal dystrophy;
9. Patients with active bleeding, bleeding tendency or unable to receive anticoagulation treatment;
10. Those with severe ventilation or ventilatory dysfunction who require continuous oxygen therapy;
11. Those who have poor compliance or cognitive impairment (such as coma, Parkinson's disease, Alzheimer's disease, drug abuse), are unable to comply with requirements or refuse to cooperate in completing study follow-up visits;
12. Other reasons causing life expectancy to be less than 1 year, such as malignant tumors and immunodeficiency diseases;
13. Other situations in which patients are not suitable for artificial aortic valve replacement or are not suitable to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Compliance rate of prosthetic valve function | 1 month following patient enrollment completion
  The compliance rate of prosthetic valve function evaluation at 1 month after surgery. The standard of prosthetic valve function is as follows: prosthetic valve pressure difference <20mmHg or peak flow rate < 3m/s, no moderate or above intravalvular regurgitation or paravalvular leakage), and no reintervention is required.
Surgery success rate | 1 month following patient enrollment completion
  Event-free survival of the prosthetic valve at 1 month postoperatively. Prosthetic valve degeneration includes stenosis and/or regurgitation due to structural abnormalities of the valve itself (e.g., leaflet tears, detachment, calcification, fibrosis, deformation of the valve frame, and fracture of the material of the connecting parts between the valve components) (referred to as structural valve degeneration), as well as dysfunction due to infective endocarditis, perivalvular leakage, valve prosthesis-patient mismatch, valve displacement, and leaflet thrombosis (referred to as nonstructural valve degeneration). Prosthetic valve degeneration usually consists of three stages, with the first stage consisting of morphological evidence of valve degeneration and structural abnormalities, before significant hemodynamic changes are evident.

SECONDARY OUTCOMES:
EOA | baseline and 1 month, 6months, 12months following patient enrollment completion
  Use echocardiography to evaluate the effective valve orifice area(EOA) to assess the hemodynamic Performance.
Mean transvalvular pressure difference | baseline and 1 month, 6months, 12months following patient enrollment completion
  Use echocardiography to measure the mean transvalvular pressure difference.
Peak flow velocity | baseline and 1 month, 6months, 12months following patient enrollment completion
  Use echocardiography to measure the peak flow velocity.
Regurgitation | baseline and 1 month, 6months, 12months following patient enrollment completion
  Evaluate the presence or absence of intravalvular or paravalvular regurgitation during the follow-up period by echocardiography.
New York Heart Association Assessment (NYHA) | baseline and 1 month, 6months, 12months following patient enrollment completion
  Evaluate New York Heart Association Assessment (NYHA) to see Heart Function Improvement.
BNP or NT-proBNP | baseline and 1 month, 12months following patient enrollment completion
  Measure BNP or NT-proBNP to get the changes in postoperative cardiac function from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No